CLINICAL TRIAL: NCT03520725
Title: Antioxidant Capacity and Vitamin A Profile in Young Adults Who Consume a Snack Bar Made From Tropical Fruits Treated With UV-C.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Investigación en Alimentación y Desarrollo A.C. (Other)
Collaborators: Universidad de Sonora (Other)
Responsible Party: Principal Investigator, Humberto Francisco Astiazaran Garcia, PhD, Principal Investigator, Centro de Investigación en Alimentación y Desarrollo A.C.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HFAG001
Record Dates: First submitted 2018-02-23; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-01

CONDITIONS: Nutritional and Metabolic Disease
Keywords: antioxidant capacity
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- No Intervention (Experimental): This group did not have an intervention
  Interventions: Other: No Intervention
- Intervention pineapple (Experimental): Daily consumption of 30 g of pineapple snack bar for 4 weeks.
  Interventions: Dietary Supplement: Pineapple snack bar
- Intervention mango (Experimental): Daily consumption of 30 g of mango snack bar for 4 weeks.
  Interventions: Dietary Supplement: Mango snack bar

INTERVENTIONS:
Other: No Intervention — This gruop did not have an intervention
  Arms: No Intervention
Dietary Supplement: Pineapple snack bar — 30 g daily of pineapple snack bar
  Arms: Intervention pineapple
Dietary Supplement: Mango snack bar — 30 g daily of mango snack bar
  Arms: Intervention mango

SUMMARY:
The objective of the present study was to evaluate the impact of a snack bar on some health indicators associated with diet (plasma antioxidant capacity, lipid profile, vitamin A profile (retinol and carotenoids)) and on the nutritional status (impact on energy and nutrients consumed) in a group of upper level students.

DETAILED DESCRIPTION:
A blind randomized controlled clinical study of healthy adults, which was carried out with the approval of the ethics committee of the Centro de Investigación en Alimentación y Desarrollo, A.C. (CIAD, A.C.) with registration CE/001/2017. The intervention was carried out in a public university in Mexico from January to April 2017. Each subject signed an informed consent form. This study lasted 30 days (4 weeks), where each participant consumed daily a snack bar irradiated with UV-C. The participants were personally interviewed by the research team with a structured selection questionnaire. Thirty subjects who met the inclusion criteria were recruited, 15 of them men and 15 women. Through a simple randomization process, the participants were assigned in 3 groups of 10 people each with 5 women and 5 men, subsequently treatments (without treatment, pineapple snack bar, or mango snack bar) were randomly assigned. The outcomes between groups were analyzed with one way ANOVA, with a P-value of 0.05 or less when there was statistical significance, using statistical software. The participants, and the laboratory technicians were blinded to the treatment assignments until the conclusion of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Young adults of 18 years of age or older,
* Healthy in appearance

Exclusion Criteria:

* People in current medical treatment
* Used antibiotics in past 15 days
* Have presented infectious symptoms on previous days
* Smokers
* Narcotic consumers
* Women in use of hormonal treatment
* Contraceptives or pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change Oxygen Radical Absorbance Capacity Assay (Antioxidant Capacity) | Change from baseline at thirty days
  From baseline and thirty days post treatment
Change Trolox Equivalent Antioxidant Capacity (Antioxidant Capacity) | Change from baseline at thirty days
  From baseline and thirty days post treatment
Change Serum Retinol Determination | Change from baseline at thirty days
  From baseline and thirty days post treatment
Change Serum pro-VA carotenoids | Change from baseline at thirty days
  From baseline and thirty days post treatment

SECONDARY OUTCOMES:
Change Serum total polyphenols determination | Change from baseline at thirty days
  From baseline and thirty days post treatment
Change Serum cholesterol determination | Change from baseline at thirty days
  From baseline and thirty days post treatment
Change Serum Triacylglycerides determination | Change from baseline at thirty days
  From baseline and thirty days post treatment
Change Serum high density lipoprotein cholesterol | Change from baseline at thirty days
  From baseline and thirty days post treatment
Change Body Mass Index | Change from baseline at thirty days
  From baseline and thirty days post treatment
Change Body composition by fat-free mass index | Change from baseline at thirty days
  From baseline and thirty days post treatment
Change Body composition by fat mass index | Change from baseline at thirty days
  From baseline and thirty days post treatment
24-hour dietary recall | Baseline and thirty days
  From baseline and thirty days post treatment

IPD SHARING:
Plan to Share IPD: No
The data base will not be shared, each collaborator will participate verifying the handling of the samples and the process of analysing the results in a blinded manner.